CLINICAL TRIAL: NCT07217210
Title: Acute Effects of a Multi-Ingredient Preworkout Supplement on Peak Torque and Muscle Activation During an Isokinetic Fatigue Protocol
Brief Title: Multi-Ingredient Preworkout Supplement on Peak Torque and Muscle Activation During Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: #HS22-0139
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male
Keywords: isometric; concentric; eccentric; leg extensors; quadriceps; electromyography

STUDY DESIGN:
Intervention Model Description: Within-subjects, placebo-controlled, crossover design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement group (Experimental): Multi-ingredient preworkout supplement
  Interventions: Dietary Supplement: Multi-ingredient preworkout supplement
- Placebo group (Placebo Comparator): Microcystalline cellulose
  Interventions: Dietary Supplement: Multi-ingredient preworkout supplement

INTERVENTIONS:
Dietary Supplement: Multi-ingredient preworkout supplement — Experimental supplement.

SUMMARY:
The primary purpose of the present study was to examine the acute effects of a MIPS product on peak torque production of the leg extensors during a fatiguing isokinetic protocol involving isometric, concentric, and eccentric muscle actions. In addition, we investigated the effects of the MIPS supplement on EMG amplitude and median power frequency (MDF) responses from the vastus lateralis, rectus femoris, and vastus medi-alis muscles.

DETAILED DESCRIPTION:
In the past several years, the use of multi-ingredient pre-workout supplements (MIPS) has become extremely popularized, and their ergogenic potential has become well-established for various sports and within the general population by both competi-tive and recreational athletes [1-6]. Some of the more prevalent ingredients in MIPS in-clude caffeine, β-alanine, L-citrulline, L-arginine, and creatine, with many of these in-gredients and others often combined into proprietary blends [7]. Although recent find-ings indicate synergistic effects among these ingredients may be present [8], it has been suggested that caffeine is the predominant factor responsible for the acute ergogenic effects associated with MIPS [2,9]. In fact, the recommended timing for ingestion of most MIPS is likely based on the stimulating effects of caffeine which typically peaks in the bloodstream 30-60 minutes post-ingestion [10,11]. As a nutritional supplement, caffeine has been shown to be beneficial for maintaining maximal strength and endur-ance as well as improving time-trial performance and other forms of high-intensity ex-ercise [10,11]. These effects have been attributed to improved motor unit firing rates and calcium release from the sarcoplasmic reticulum, subsequently enhancing muscle contraction force [4,12]. β-alanine is another ingredient included in most MIPS [7] and has been identified as the rate-limiting precursor to carnosine, an intracellular muscle buffer [13]. Supplementation with β-alanine has been shown to increase intramuscular levels of carnosine, thereby attenuating metabolic acidosis during high-intensity exer-cise [13]. As precursors to the potent vasodilator, nitric oxide, both L-citrulline and L-arginine supplements have been demonstrated to enhance blood flow to active mus-cles, subsequently delaying the onset of muscular fatigue [14-16]. Based on these collec-tive physiological mechanisms, a MIPS containing these notable ergogenic ingredients (caffeine, β-alanine, L-citrulline, L-arginine) may provide neuromuscular benefits for sustaining force or power output during various forms of vigorous activity.

The vast majority of previous investigations examining the acute effects of MIPS on performance have focused on isotonic variables of upper and lower body muscular strength [i.e. bench press, leg press, and squat one-repetition maximum (1-RM), maxi-mum voluntary contractions (MVC)], endurance (i.e. repetitions to failure at %1-RM), and power (vertical jump, Wingate Anaerobic testing, and critical power) [1-6,9,12,18,19]. Despite conflicting evidence for maximal force and power production [4,6,20,21], the findings of several studies [1,3,4,12,17-19,22,23] have largely indicated acute MIPS supplementation can enhance overall force retention and muscular endur-ance during prolonged or intermittent bouts of high intensity activity. Currently, how-ever, the exact underlying mechanisms responsible for these benefits on neuromuscular function are poorly understood.

Isokinetic dynamometers coupled with surface electromyography (EMG) record-ings are two frequently utilized instruments for the non-invasive assessment of neu-romuscular function and fatigue during static and dynamic muscle actions [24-27]. The utility of isokinetic testing involves the ability to measure isometric, concentric, and eccentric torque levels across an entire range of motion at controlled velocities with minimal skill involvement required. Results from isokinetic testing can provide torque production at different joint angles, while identifying muscle imbalances, tracking the recovery process from injury or surgery, and measuring the rate of force development [28,29]. Thus, as both a training and assessment tool, isokinetic testing is common in clinical and performance settings.

Surface electromyography (EMG) is a technique that involves recording and quantifying the action potentials associated with contracting skeletal muscle fibers [30]. The amplitude contents of the EMG signal reflect the level of muscle activation (i.e. motor unit recruitment and firing rates) [31], whereas the frequency contents pro-vide information related to the muscle fiber conduction velocity [32]. To our knowledge, only one study [5] has directly examined EMG responses associated with acute MIPS administration. Specifically, Negro et al. [5] reported acute MIPS (creatine, arginine, β-alanine, glutamine, taurine) ingestion improved EMG-based indicators of fatigue (i.e. conduction velocity, fractal dimension) during sustained isometric contrac-tions following a resistance exercise protocol designed to elicit fatigue. The authors [5] proposed these acute benefits of their MIPS product may be attributable to improved: 1) peripheral components of performance fatiguability, 2) buffering capacity of the mus-cle from β-alanine, and 3) regulation of mechanisms associated with exercise-induced fatigue from arginine, glutamine, and taurine. Based on these findings [5], valuable in-sight can be gained into the underlying neuromuscular factors associated with MIPS ingestion by examining muscle function and fatigue through isokinetic and EMG as-sessments. Thus, the primary purpose of the present study was to examine the acute ef-fects of a MIPS product on peak torque production of the leg extensors during a fatigu-ing isokinetic protocol involving isometric, concentric, and eccentric muscle actions. In addition, we investigated the effects of the MIPS supplement on EMG amplitude and median power frequency (MDF) responses from the vastus lateralis, rectus femoris, and vastus medialis muscles.

ELIGIBILITY:
Inclusion Criteria:

* Male, 19-29 years of age, one year of resistance training experience

Exclusion Criteria:

* Subjects were eligible to participate if they did not report: 1) cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders; 2) use of any medications; 3) use of nutritional supplements; 4) habitual use of caffeine (≥ 1 caffeinated beverage per day); or 5) participation in another clinical trial or investigation of another nutritional product within 30 days of screening/enrollment.

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Peak torque | Two days.
  Isometric, concentric, and eccentric.

SECONDARY OUTCOMES:
EMG responses. | 60 minutes per visit over the course of two visits (each separated by one week).
  Relative amplitude and median power frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Camic, PHD, Principal Investigator — Northern Illinois University
Locations (1):
- Northern Illinois University, DeKalb, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The informed consent and IRB application indicated that individual data would not be shared.